CLINICAL TRIAL: NCT03039530
Title: Impact of Public Health Nurse Delivered Group CBT for Postpartum Depression on Women and Their Children: A Randomized Controlled Trial
Brief Title: Group CBT for PPD in the Public Health Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Niagara Region Public Health (Other)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, Assistant Professor, Department of Psychiatry and Behavioural Neurosciences, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PH CBT
Record Dates: First submitted 2017-01-19; First posted 2017-02-01 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Depression, Postpartum
Keywords: Postpartum Depression; Cognitive Behavioral Therapy; Public Health; Mother; Infant; Emotion
MeSH Terms: conditions — Depression, Postpartum | interventions — Postnatal Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Group CBT for PPD. Women in the treatment group will attend a 9-week group CBT intervention for PPD. This intervention was developed at the Women's Health Concerns Clinic (WHCC) at St. Joseph's Healthcare Hamilton. It was designed to be brief, simple, and applicable to women in community settings. It consists of 9 weekly 2-hour sessions where core CBT skills are learned and practiced, and a new psychoeducational topic is introduced and discussed by women each week.
  Interventions: Behavioral: Group Cognitive Behavioral Therapy
- Control Group (Active Comparator): Standard Care. The usual care group will receive standard care from their family physician and midwife or obstetrician. They will also be made aware of the perinatal programming available to them through Niagara Region Public Health. Women and family physicians will also receive a copy of the Canadian Practice Guidelines for the Treatment of Perinatal Depression.
  Interventions: Behavioral: Postnatal Care As Usual

INTERVENTIONS:
Behavioral: Group Cognitive Behavioral Therapy — 9 weekly 2-hour group CBT sessions delivered by 2 trained Public Health Nurses.
  Arms: Treatment Group
Behavioral: Postnatal Care As Usual — Postnatal care as usual will involve treatment from their family physician and midwife or obstetrician, and voluntary participation in programs offered by Niagara Region Public Health and in the community.
  Arms: Control Group

SUMMARY:
Postpartum depression (PPD) affects over 14,000 women in Ontario each year and can have profound effects on mothers, their children, and their families. The cost of one case of PPD exceeds $150,000, a significant proportion of which is related to its impact on offspring. However, difficulties accessing preferred treatments (e.g., psychotherapy) result in fewer than 15% of women receiving care. While Public Health Units have played an important role in PPD detection in Ontario, Public Health Nurses (PHNs) currently lack the skills to deliver evidence-based treatment to women. Cognitive Behavioural Therapy (CBT) delivered in group format is effective for treating depression in the perinatal period, and as PHNs are often the first point of contact for women experiencing PPD, with specialized training it is likely that they can deliver high-quality CBT.

The primary objective of this study is to determine if PHNs can be trained to deliver group Cognitive Behavioral Therapy (CBT) to acutely treat PPD, reduce relapse and recurrence, improve mother-infant attachment and parenting and optimize infant emotional functioning.

DETAILED DESCRIPTION:
In addition to its effects on maternal health, PPD can adversely affect mother-infant attachment, parenting, and the development and health of her children. The negative effects of PPD on offspring can include an increased risk of insecure attachment, poorer cognitive, language, and behavioral development, as well as an increased risk of emotion regulatory problems. To determine if PHNs can effectively deliver group CBT for PPD that is superior to postnatal care as usual, the investigators will proceed with a randomized controlled trial (RCT). Women in the treatment group will attend a 9-week group CBT intervention delivered by trained PHNs. Those in the control group will receive standard postnatal care.

This RCT will compare the effects of group CBT to postnatal care as usual on maternal depression, anxiety, mother-infant attachment, parenting, healthcare utilization and social support, as well as infant development, emotion regulation, and healthcare utilization

ELIGIBILITY:
Inclusion Criteria:

* Eligible women will be >18 years of age, understand and speak English (so that they can participate in the CBT group and complete study measures), have an EPDS score between 10 and 23. They will also all be within 12 months of delivering an infant

Exclusion Criteria:

* Women can have psychiatric comorbidities with the exception of bipolar disorder, a current psychotic, substance or alcohol use disorder, or antisocial or borderline personality disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | 6 months
  The EPDS will be used to assess maternal depression. A score of >12 is consistent with PPD and changes in scores >4 are indicative of clinically significant improvement.
Mini International Neuropsychiatric Interview - Current Major Depressive Disorder | 6 months
  Used to assess maternal depression.

SECONDARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) | 6 months
  Maternal Anxiety will be assessed using the Penn State Worry Questionnaire.
Postpartum Bonding Questionnaire | 6 months
  Used to detect disorders of the mother-infant relationship.
Parent-Child Early Relational Assessment | 6 months
  Used to measure the quality of affect and behavior in parent-child interactions.
Social Provisions Scale | 6 months
  Used to measure the degree to which mothers' social relationships provide support
Ages and Stages Questionnaires - Third Edition | 6 months
  Assesses infant communication, motor and socioemotional development using age-specific scales.
Maternal & Infant Healthcare Utilization | 6 months
  Adopted form the Canadian Community Health Survey to track use of healthcare services.
Infant Behaviour Questionnaire-Revised | 6 months
  This scale assesses infant temperament
Face-to-Face Still Face Paradigm | 6 months
  Experimental task used to assess emotion regulation in infants
Parasympathetic Nervous System Functioning: Heart Rate Variability | 6 months
  Used to asses the flexibility of the central and peripheral nervous system to handle stress.
Salivary Cortisol | 6 months
  Used to assess stress reactivity and emotion regulation. Three samples will be taken during each assessment: 10-15 minutes after the beginning of the assessment, 15-20 minutes after the face-to-face still face task and at the end of the visit.
Corticolimbic Brain Function: EEG-Based Frontal Lobe Asymmetry (via MUSE Headband) | 6 months
  Corticolimbic brain activity at the scalp will be assessed using electroencephalography (EEG). Greater left frontal asymmetry (greater activity in the left frontal hemisphere) is thought to reflect positive emotionality and indicate a greater tendency to engage in more adaptive emotion regulation strategies. However greater right activity reflects a tendency to engage in withdrawn behaviours and negative emotionality.

CONTACTS AND LOCATIONS:
Locations (1):
- Niagara Region Public Health, Thorold, Ontario, Canada

REFERENCES:
- [Derived] Van Lieshout RJ, Layton H, Savoy CD, Haber E, Feller A, Biscaro A, Bieling PJ, Ferro MA. Public Health Nurse-delivered Group Cognitive Behavioural Therapy for Postpartum Depression: A Randomized Controlled Trial. Can J Psychiatry. 2022 Jun;67(6):432-440. doi: 10.1177/07067437221074426. Epub 2022 Jan 21. PMID 35060398